CLINICAL TRIAL: NCT05477069
Title: Feasibility Study of an Innovative Medical Device for Sampling the Contents of the Small Intestine. Functional Evaluation on the Transit of Healthy Volunteers. A First in Man, Prospective, Monocentric, Not Randomized Study.
Brief Title: Feasibility Study of an Innovative Medical Device for Sampling the Contents of the Small Intestine.
Acronym: DIGEST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Clinical Investigation Centre for Innovative Technology Network (Network); Pelican Health (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 38RC18.011
Record Dates: First submitted 2022-06-17; First posted 2022-07-28 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2023-12

CONDITIONS: Healthy Volunteers
Keywords: Innovative medical device; Microbiota; Biochemically controlled capsule; Intestinal fluid sampling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- First intervention group (Experimental): The volunteer ingests the medical device which passes through the body for a period of 12 to 24 hours. Capsules are collected and analysis on intestinal fluid and faeces are performed
  Interventions: Device: Innovative medical device for sampling small intestine content

INTERVENTIONS:
Device: Innovative medical device for sampling small intestine content — Ingestion of the medical device by the volunteer

SUMMARY:
For the first time in the world, the objective of this study is to evaluate on healthy volunteers, an innovative medical device for the capture of intestinal liquid.This medical device is not yet CE marked.

DETAILED DESCRIPTION:
This medical device consists of a standard pill made of 3 capsules for the collection of intestinal microbiota. The pill is ingested by the volunteer and multi-omics analysis will be performed on intestinal fluid samples from the capsules and also on faeces.

First in man, involving a medical device, prospective, monocentric, not randomized, not controlled and open-label study.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand the study and the associated instructions
* Aged ≥18 years and ≤65 years
* Fasting with water and food for at least 10 hours
* BMI between ≥20 and ≤30 kg/m².
* Transit evaluated at 1 to 3 bowel movements/day
* Maintain regular physical activity and eating habits for the duration of the study
* Affiliated with a social security plan
* Have a freezer in their home and at work, if applicable
* Volunteer staying in the Isère department during the collection of the faeces (from 96 hours to 15 days max)
* Having signed the informed and collection consent

Exclusion Criteria:

Subject :

* with medical treatment (except oral contraception and/or probiotics and related products)
* with lactose and fructose intolerance
* with of gastroparesis
* who had a colonoscopy preparation up to 1 month prior to inclusion
* in the exclusion period of another clinical investigation,
* who receive more than 4500 euros of compensation due to his participation in other biomedical research in the 12 months preceding this study
* who cannot be contacted in case of emergency
* who has taken during the 15 days prior to inclusion and/or is scheduled to take the following treatments during the study: antidepressants, anxiolytics, antiparkinsonian agents, neuroleptics, antibiotics and prebiotics
* who has taken during the previous 7 days: at least once a treatment for irritable bowel syndrome (antispasmodics,..) or for constipation (laxative) or for diarrhea
* with a known food allergy
* who have to undergo colon surgery
* with intestinal obstruction history
* with hepatic, cardiac, congenital or renal comorbidity
* with long-standing diabetes
* with an inflammatory disease of the digestive tract, a history of digestive surgery
* who have been treated with radiotherapy or who have taken anti-inflammatory drugs for a long time
* with gastric fullness
* with known or suspected obstruction of the gastrointestinal tract (including known inflammatory bowel or intestinal diverticula)
* with presence of swallowing disorders or Zencker's diverticulum
* with nausea, deviated nasal septum
* with contraindications to esophageal tube placement (chronic esophageal pathology)
* drug or alcohol abuse (3 units for men and 2 units for women according to WHO criteria)
* with a known allergy to silicone or to iodine
* refusing medical imaging or surgery (in case of non-recovery of the capsule)
* protected person concerned by the articles L1121-5 to L1121-8 of the Public Health Code
* absence of highly effective contraception for women with childbearing capacity until the end of the cycle following the end of participation in the trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-10-24 (Actual); Primary Completion 2023-11-06 (Actual); Study Completion 2023-11-06 (Actual)

PRIMARY OUTCOMES:
Demonstrate the absence of adverse events (safety of the medical device) and that the device is analyzable (performance of the medical device). | From 96 hours to 15 days
  Safety is assessed with the absence of grade >3 adverse events. Performance is assessed by the presence of at least one capsule found in the stool with a satisfactory visual condition of capsule and with a sufficient volume of its contents within 96 hours after ingestion.
  The primary objective of this study is met if safety and performance are achieved for at least 12 of 15 volunteers.

SECONDARY OUTCOMES:
Number and grade of adverse events collected during the capsule collection period | From 96 hours to 15 days
  In order to verify the safe use of the medical device the number and grade of adverve events are collected from 96 hours to 1 month.
Number of capsules found to verify that the medical device passes through the human body | From 96 hours to 15 days
  Recovery of 3 capsules per volunteer
Verify that the medical device has captured intestinal fluid | From 96 hours to 15 days
  Measurement of the volume contained in each capsule.
Verify that the medical device has opened in the intestine | From 96 hours to 15 days
  pH measurement of the contents of each capsule.
Absence of tears and detachment of the various elements of the capsule | From 96 hours to 15 days
  Visual inspection of the capsule after collection to determine absence of tears and detachment of the various elements
Metagenomic analysis using 16s sequencing will provide data to establish differences in the gut microbiota profile/composition between capsule and faecal contents. | From 96 hours to 15 days
  Metabolomic profile of capsule and faecal contents will be assessed by untargeted metabolomics. Identification, relative quantification and listing of metabolites specific to a sampling method will be generated.Microbiota will be described in terms of alpha and beta diversity, phylum, genus, OTU
Medical device usability and acceptability : descriptive analysis | From 96 hours to 15 days
  Registration of volunteer sensation during medical device ingestion using a questionnaire without scale. A descriptive analysis will be done with the answers.
Obtain an overview of the sample's functional potential and identify biomarkers (organisms) via culturomics, on samples from up to 2 subjects. | From 96 hours to 2 months
  Results of culturomic analysis of capsule contents, on up to 2 subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Matthieu, MD, PhD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- University Hospital Grenoble Alpes, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tronel A, Silvent AS, Buelow E, Giai J, Leroy C, Proust M, Martin D, Le Gouellec A, Soranzo T, Mathieu N. Pilot Study: Safety and Performance Validation of an Ingestible Medical Device for Collecting Small Intestinal Liquid in Healthy Volunteers. Methods Protoc. 2024 Feb 4;7(1):15. doi: 10.3390/mps7010015. PMID 38392689
- [Derived] Tronel A, Roger-Margueritat M, Plazy C, Cunin V, Mohanty I, Dorrestein PC, Soranzo T, Le Gouellec A. Untargeted and semi-targeted metabolomics approach for profiling small intestinal and fecal metabolome using high-resolution mass spectrometry. Metabolomics. 2025 Jun 19;21(4):84. doi: 10.1007/s11306-025-02288-2. PMID 40537703